CLINICAL TRIAL: NCT04663347
Title: A Phase 1b/2, Open-Label Trial to Assess the Safety and Preliminary Efficacy of Epcoritamab (GEN3013; DuoBody®-CD3xCD20) in Combination With Other Agents in Subjects With B-cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: Safety and Efficacy Trial of Epcoritamab Combinations in Subjects With B-cell Non-Hodgkin Lymphoma (B-NHL)
Acronym: EPCORE™ NHL-2
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT3013-02; 2023-504805-35-00 (EU CTIS Number); 2020-000845-15 (EudraCT Number); NL74222.056.20 (Registry Identifier: CCMO); 283235 (Other: IRAS ID; UK Research Summaries Database); RECF4377 (Other: The French National Cancer Institute)
Expanded Access: NCT05733650 (Approved for marketing)
Record Dates: First submitted 2020-10-27; First posted 2020-12-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma; Follicular Lymphoma
Keywords: DuoBody®; monoclonal antibodies; anti-CD3; anti-CD20
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; R-CHOP protocol; Lenalidomide; Bendamustine Hydrochloride; Cytarabine; Dexamethasone; Oxaliplatin; Carboplatin; Gemcitabine; Ifosfamide; etoposide phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Arm 1 - Epcoritamab + R-CHOP (Experimental): In participants with previously untreated DLBCL.
  Interventions: Drug: rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone; Biological: Epcoritamab
- Arm 2 - Epcoritamab + R2 (Experimental): In participants with R/R FL.
  Interventions: Biological: Epcoritamab; Drug: Rituximab and Lenalidomide
- Arm 3 - Epcoritamab + BR (Experimental): In participants with previously untreated FL.
  Interventions: Drug: rituximab and bendamustine; Biological: Epcoritamab
- Arm 4 - Epcoritamab + R-DHAX/C (Experimental): In participants with R/R DLBCL eligible for ASCT.
  Interventions: Drug: rituximab, cytarabine, dexamethasone, and oxaliplatin/carboplatin; Biological: Epcoritamab
- Arm 5 - Epcoritamab + GemOx (Experimental): In participants with R/R DLBCL ineligible ASCT.
  Interventions: Drug: gemcitabine and oxaliplatin; Biological: Epcoritamab
- Arm 6 - Epcoritamab + R2 (Experimental): In participants with previously untreated FL.
  Interventions: Drug: rituximab and lenalidomide; Biological: Epcoritamab
- Arm 7 - Epcoritamab maintenance (Experimental): In participants with FL who achieved a CR or PR after receiving SOC treatment in 1L or 2L.
  Interventions: Biological: Epcoritamab
- Arm 8 - Epcoritamab + R mini-CHOP (Experimental): In participants with previously untreated DLBCL who are ineligible to receive full-dose anthracycline.
  Interventions: Drug: rituximab, cyclophosphamide, reduced dose of doxorubicin, vincristine, and prednisone; Biological: Epcoritamab
- Arm 9 - Epcoritamab + Lenalidomide (Experimental): In participants with R/R FL who progressed within 24 months of initiation of first-line anti-CD20-containing immunochemotherapy.
  Interventions: Drug: Lenalidomide; Biological: Epcoritamab
- Arm 10 - Epcoritamab + R-ICE (Experimental): In participants with R/R DLBCL eligible for ASCT.
  Interventions: Drug: rituximab, ifosfamide, carboplatin, and etoposide phosphate; Biological: Epcoritamab

INTERVENTIONS:
Drug: rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone — 6 cycles (21-day cycles)
  Other Names: R-CHOP
  Arms: Arm 1 - Epcoritamab + R-CHOP
Drug: rituximab and lenalidomide — rituximab 6 cycles and lenalidomide 12 cycles (28-day cycles)
  Other Names: R2
  Arms: Arm 6 - Epcoritamab + R2
Drug: rituximab and bendamustine — 6 cycles (28-day cycles)
  Other Names: BR
  Arms: Arm 3 - Epcoritamab + BR
Drug: rituximab, cytarabine, dexamethasone, and oxaliplatin/carboplatin — 3 cycles (21-day cycles)
  Other Names: R-DHAX/C
  Arms: Arm 4 - Epcoritamab + R-DHAX/C
Drug: gemcitabine and oxaliplatin — 4 cycles (28-day cycles)
  Other Names: GemOx
  Arms: Arm 5 - Epcoritamab + GemOx
Biological: Epcoritamab — Every week in cycle 1-4, every 3 weeks in cycle 5 and 6, followed by every 4 weeks in cycle 7 for a total of 1 year.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 1 - Epcoritamab + R-CHOP
Drug: rituximab, cyclophosphamide, reduced dose of doxorubicin, vincristine, and prednisone — 6 cycles (21-day cycles)
  Other Names: R mini-CHOP
  Arms: Arm 8 - Epcoritamab + R mini-CHOP
Drug: Lenalidomide — 12 cycles (28-day cycles)
  Arms: Arm 9 - Epcoritamab + Lenalidomide
Drug: rituximab, ifosfamide, carboplatin, and etoposide phosphate — 3 cycles (21-day cycles)
  Other Names: R-ICE
  Arms: Arm 10 - Epcoritamab + R-ICE
Biological: Epcoritamab — Every week in cycle 1-3, every 2 weeks in cycle 4-9, followed by every 4 weeks for a total of 2 years.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 3 - Epcoritamab + BR
Biological: Epcoritamab — Every week in cycle 1 and 2, followed by every 4 weeks for a total of 2 years.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 6 - Epcoritamab + R2
Biological: Epcoritamab — Every week in cycle 1 and then every 8 weeks for a total of 2 years.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 7 - Epcoritamab maintenance
Biological: Epcoritamab — Every week in cycles 1 and 2, then every 3 weeks in cycles 3 to 6 and then every 4 weeks for cycles 7 and 8.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 8 - Epcoritamab + R mini-CHOP
Biological: Epcoritamab — Every week in cycle 1-3 and then every 4 weeks for a total of 2 years.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 9 - Epcoritamab + Lenalidomide
Biological: Epcoritamab — Every week in cycle 1-4, every 2 weeks in cycle 5-9 followed by every 4 weeks until ASCT or disease progression.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 10 - Epcoritamab + R-ICE; Arm 4 - Epcoritamab + R-DHAX/C
Biological: Epcoritamab — Eligible participants will receive subcutaneous (SC) epcoritamab in 28-day cycles. Fixed-treatment epcoritamab will be administered following a 2-Set Up Dosing regimen in Cycle 1. There will be 2 cohorts, 2a and 2b with different dosing schedules.
  Cohort 2a will be dosed weekly (QW) in Cycles 1-3, once every 2 weeks (Q2W) in Cycles 4-9, and once every 4 weeks (Q4W) in Cycle 10 and beyond for up to 2 years.
  In cohort 2b, an alternate dosing schedule for epcoritamab will be explored: epcoritamab administered QW for Cycles 1-2 only, then Q4W in Cycle 3 and beyond for up to 2 years.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 2 - Epcoritamab + R2
Drug: Rituximab and Lenalidomide — Rituximab 375 milligrams per meter squared (mg/m^2) will be administered intravenously QW in Cycle 1 and Q4W in Cycles 2-5. Lenalidomide 20 mg will be administered orally daily for 21 days for 12 cycles.
  Other Names: R2
  Arms: Arm 2 - Epcoritamab + R2
Biological: Epcoritamab — Cycle 1-3 every week, every other week Cycle 4-9 and then Q4W until progression or unacceptable toxicity.
  Other Names: GEN3013; DuoBody®-CD3xCD20; EPKINLY™
  Arms: Arm 5 - Epcoritamab + GemOx

SUMMARY:
The purpose of this trial is to measure the safety and effectiveness of epcoritamab (EPKINLY™), either by itself or together with other therapies, when treating participants with B-cell non-Hodgkin Lymphoma (B-NHL). The aim of the first part of the trial is to identify the most appropriate dose of epcoritamab, and the aim of the second part of the trial is to assess the selected epcoritamab dose in a larger group of participants with B-NHL. All participants in this trial will receive either epcoritamab alone, or epcoritamab combined with another standard treatment regimen, with a total of 10 different treatment arms being studied.

Trial details include:

* The treatment duration for each participant depends upon which arm of treatment they are assigned to.
* The visit frequency for each participant depends upon which arm of treatment they are assigned to, but will be weekly to start for all participants, then will decrease to either: every 2 weeks, or every 3 weeks, or every 4 weeks, or every 8 weeks.
* All participants will receive active drug; no one will be given placebo.

Participants who receive treatment with epcoritamab will have it injected right under the skin. Participants will receive a different regimen of epcoritamab depending upon which arm of treatment they are assigned.

Participants who receive standard treatments will have intravenous (IV) infusions and/or oral administration of those treatments. Participants will receive a different standard treatment regimen depending upon which arm of treatment they are assigned.

DETAILED DESCRIPTION:
A Phase 1b/2, open-label, multinational, interventional trial to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics/biomarkers, immunogenicity, and preliminary efficacy of epcoritamab in combination with other standard of care (SOC) agents in participants with B-NHL.

All participants in the trial will receive epcoritamab, as monotherapy or in combination. The following regimens will be investigated:

* Arm 1: epcoritamab + rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in participants with previously untreated diffuse large B-cell lymphoma (DLBCL)
* Arm 2: epcoritamab + rituximab and lenalidomide (R2) in participants with relapsed/refractory (R/R) follicular lymphoma (FL)
* Arm 3: epcoritamab + rituximab and bendamustine (BR) in participants with previously untreated FL
* Arm 4: epcoritamab + rituximab, cytarabine, dexamethasone, and oxaliplatin/ carboplatin (R-DHAX/C) in participants with R/R DLBCL eligible for autologous stem cell transplant (ASCT)
* Arm 5: epcoritamab + gemcitabine and oxaliplatin (GemOx) in participants with R/R DLBCL ineligible for ASCT due to age, performance status (PS), or comorbidity
* Arm 6: epcoritamab + R2 in participants with previously untreated FL
* Arm 7: epcoritamab maintenance in participants with FL who achieve a complete response (CR) or a partial response (PR) following first or second line SOC treatment
* Arm 8: epcoritamab + reduced dose of R-CHOP (R mini-CHOP) in participants with previously untreated DLBCL who are ineligible to receive full-dose anthracycline
* Arm 9: epcoritamab + lenalidomide for second-line treatment in participants with R/R FL who progressed within 24 months of initiation of first-line anti-CD20-containing immunochemotherapy
* Arm 10: epcoritamab + rituximab, ifosfamide, carboplatin, and etoposide phosphate (R-ICE) in participants with R/R DLBCL eligible for ASCT

The trial consists of two parts: Part 1 ('Dose Escalation') and Part 2 ('Dose Expansion'). The primary objective of Part 1 is safety, and it includes Arm 1-5 and Arm 10. Part 2 includes all 10 arms (Arm 1-10) and the primary goal of all arms, except Arm 7, is preliminary efficacy. For Arm 7, the primary goal is safety. Participants in Arm 1-5 and Arm 10 can only participate in either Part 1 or Part 2. Dose Limiting Toxicities (DLTs) will be assessed in Part 1 and for a selected number of participants in Arm 8 during a 28-day period (safety run-in). The arms are conducted in parallel.

ELIGIBILITY:
Key Inclusion Criteria

1. Measurable disease defined as ≥1 measurable nodal lesion (long axis >1.5 cm and short axis >1.0 cm) or ≥1 measurable extra-nodal lesion (long axis >1.0 cm) on computed tomography (CT) or magnetic resonance imaging (MRI). Applies to all arms except arm 7.
2. Eastern Cooperative Oncology Group (ECOG) PS score of 0, 1 or 2
3. Acceptable organ function at screening
4. CD20-positive non-Hodgkin lymphoma (NHL) at most recent representative tumor biopsy
5. If of childbearing potential participant must practicing a highly effective method of birth control
6. A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control

Arm 1:

* Newly diagnosed DLBCL
* DLBCL, not otherwise specified (NOS)
* "Double-hit" or "triple-hit" DLBCL
* FL Grade 3B

Arm 2: R/R FL

Arm 3: Newly diagnosed, previously untreated FL grade 1-3A

Arm 4:

* Documented R/R DLBCL and eligible for HDT-ASCT
* DLBCL, NOS
* "Double-hit" or "triple-hit" DLBCL
* FL Grade 3B

Arm 5:

* Documented R/R DLBCL and ineligible for HDT-ASCT
* DLBCL, NOS
* "Double-hit" or "triple-hit" DLBCL
* FL Grade 3B

Arm 6: Newly diagnosed, previously untreated FL grade 1-3A

Arm 7:

* FL Grade 1-3A
* If PR or CR per Lugano criteria following first-line or second-line treatment with SOC regimen, and last dose of SOC within 6 months prior to enrollment.

Arm 8:

* Newly diagnosed DLBCL who are not fit to receive full-dose anthracycline
* T-cell/histiocyte rich DLBCL
* "Double-hit" or "triple-hit" DLBCL
* FL Grade 3B

Arm 9:

* R/R FL
* Progressed within 24 months of initiating first-line treatment

Arm 10:

* Documented R/R DLBCL and eligible for HDT-ASCT
* DLBCL, NOS
* "Double-hit" or "triple-hit" DLBCL
* FL Grade 3B

Key Exclusion Criteria

1. Chemotherapy, radiation therapy, or major surgery within 4 weeks prior to the first dose of epcoritamab
2. Any prior treatment with a bispecific antibody targeting CD3 and CD20.
3. Treatment with CAR-T therapy within 100 days prior to first dose of epcoritamab
4. Clinically significant cardiovascular disease
5. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
6. CNS lymphoma or known CNS involvement by lymphoma at screening as confirmed by MRI/CT scan of the brain and, if clinically indicated, by lumbar puncture
7. Positive tests for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
8. Known history of seropositivity of human immunodeficiency virus (HIV)
9. Active tuberculosis or history of completed treatment for active tuberculosis within the past 12 months
10. Neuropathy > grade 1
11. Receiving immunostimulatory agent
12. Prior allogeneic HSCT
13. Current seizure disorder requiring anti-epileptic therapy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Dose limiting Toxicities (DLTs) | During the first cycle (Cycle length= 28 days) in each cohort
  DLT events are defined as clinically significant adverse events (AEs) or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications as assessed per Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria version 5.0.
Part 1 and Part 2 (Arms 1-5, 7 and 10): Number of Participants With Adverse Events (AEs) | From first dose of drug until either 60 days after last dose, date participant withdraws consent, date participant starts a new systemic anticancer therapy, or date participant dies, whichever occurs first (up to approximately 3 years)
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign. (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Part 2 (Except Arm 7): Overall Response Rate (ORR) | Up to 3 years
  ORR is defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on Lugano criteria.

SECONDARY OUTCOMES:
Part 1 and 2: Clearance (CL) of Epcoritamab | Predose and postdose at multiple timepoints until treatment discontinuation (up to 3 years)
Part 1 and 2: Area Under the Concentration-Time Curve (AUC) of Epcoritamab | Predose and postdose at multiple timepoints until treatment discontinuation (up to 3 years)
Part 1 and 2: Maximum (Peak) Plasma Concentration (Cmax) of Epcoritamab | Predose and postdose at multiple timepoints until treatment discontinuation (up to 3 years)
Part 1 and 2: Time to Reach Cmax (Tmax) of Epcoritamab | Predose and postdose at multiple timepoints until treatment discontinuation (up to 3 years)
Part 1 and 2: Terminal Elimination Half-Life (t 1/2) of Epcoritamab | Predose and postdose at multiple timepoints until treatment discontinuation (up to 3 years)
Part 1 and 2: Number of Immune Cell Populations | Up to 2 years
  Immune cell populations in peripheral blood and tumor biopsies will be assessed.
Part 1 and 2: Percentage of Immune Cell Populations | Up to 2 years
  Immune cell populations in peripheral blood and tumor biopsies will be assessed.
Part 1 and 2: Change From Baseline in Cytokine Levels up to Cycle 3 | Up to Cycle 3 (cycle length = 21 days for Arms 1, 4, 8 and 10; cycle length = 28 days for Arms 2, 3, 5, 6 and 9; cycle length = 28 days (Cycle 1) and 56 days (Cycles 2, 3) for Arm 7)
  Change in cytokine levels in peripheral blood samples will be assessed.
Part 1 and 2: Change From Baseline in Circulating Tumor Deoxyribonucleic Acid (DNA) Level up to End of Treatment (up to 2 Years) | Up to 2 years
  Change in circulating tumor DNA levels will be assessed.
Part 1 and 2: Number of Participants With Anti-Drug Antibodies (ADAs) to Epcoritamab | Up to 3 years
Part 1: ORR | Up to 3 years
  ORR is defined as the percentage of participants achieving CR or PR based on Lugano criteria.
Part 1 and 2: Duration of Response (DOR) | Up to 3 years
  DOR: the time from the first documentation of objective tumor response (CR or PR) to the date of first PD or death, whichever occurs earlier, based on Lugano criteria.
Part 1 and 2: Time to Response (TTR) | Up to 3 years
  TTR is defined as the time from Day 1 of Cycle 1 to first documentation of objective tumor response (CR or PR).
Part 1 and 2: Progression Free Survival (PFS) | Up to 3 years
  PFS is defined as the time from Day 1 of Cycle 1 to first documented PD or death due to any cause, whichever occurs earlier, based on Lugano criteria.
Part 1 and 2: Overall Survival (OS) | Up to 3 years
  OS is defined as the time from the date of first dose, to the date of death due to any cause.
Part 1 and 2: Time to Next Anti-lymphoma Therapy (TTNT) | Up to 3 years
  TTNT is defined as the time from Day 1 of Cycle 1 to first documented administration of subsequent anti-lymphoma therapy.
Part 1 and 2: Percentage of Participants With Minimal Residual Disease (MRD) Negativity | Up to 3 years
  It is defined as the percentage of participants with at least 1 MRD negative result.
Part 1 and 2: Duration of minimal residual disease (MRD) negativity | Up to 3 years
Part 2 (Arm 7): Percentage of Participants Who Converted From MRD Positivity to MRD Negativity | Up to 3 years
Part 2 (Except Arm 7): Percentage of Participants with Complete Response (CR) in Arms 1 to 10 | Up to 3 years
Part 2 (Arm 7): Percentage of Participants With CR | Week 24, Week 48, and Week 96
  It is defined as the percentage of participants who remain in complete remission or converting to complete remission after first trial drug administration.
Part 1 and 2: Time to Complete Response (TTCR) | Up to 3 years
  TTCR is defined as the time from first trial drug administration to the date of first documented complete response post-treatment.
Part 1 and 2: Duration of Complete Response (DoCR) | Up to 3 years
  DoCR is defined as the time from the first documentation of CR to the date of PD or death, whichever occurs first based on Lugano criteria.
Part 2: Number of Participants with AEs (Except Arm 7) | From first dose of drug until either 60 days after last dose, date participant withdraws consent, date participant starts a new systemic anticancer therapy, or date participant dies, whichever occurs first (up to approximately 3 years)
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign. (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine, Ann Arbor, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering CC, New York, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - Austin Health, Heidelberg
  - Linear Clinical Research Limited, Nedlands
- Belgium (3):
  - AZ Sint-Jan, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - CHU UCL Namur Site Godinne, Yvoir
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice v Motole, Prague
  - Vseobecna Fakultni Nemocnice, Prague
- Denmark (4):
  - Århus Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Vejle Sygehus, Vejle
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - HUS Cancer Center, Lahti
- France (4):
  - Hopital Claude Huriez - CHRU Lille, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Italy (7):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Fondazione del Piemonte per l Oncologia Istituto di Candiolo IRCCS, Candiolo
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST, Meldola
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
- Netherlands (6):
  - Amsterdam UMC, Locatie VUMC, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht, Utrecht
- Oslo Universitetssykehus HF, Radiumhospitalet, Oslo, Norway
- Spain (5):
  - ICO l Hospitalet, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Sweden (5):
  - Södra Älvsborgs Sjukhus, Borås
  - Sahlgrenska Sjukhuset, Gothenburg
  - Skånes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset, Solna
  - Akademiska Sjukhuset, Uppsala
- United Kingdom (3):
  - The Christie Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchi L, Sureda A, Leppa S, Vermaat JSP, Nijland M, Christensen JH, de Vos S, Holte H, Merryman RW, Lugtenburg PJ, Abrisqueta P, Linton KM, Sunkersett G, Hoehn D, Rana A, Abbas A, Marek J, Hao Y, Steele AJ, Morehouse C, Hutchings M, Belada D. Fixed-duration epcoritamab plus R2 drives favorable outcomes in relapsed or refractory follicular lymphoma. Blood. 2025 Nov 27;146(22):2629-2640. doi: 10.1182/blood.2025029909. PMID 40920572
- [Derived] Brody JD, Jorgensen J, Belada D, Costello R, Trneny M, Vitolo U, Lewis DJ, Karimi YH, Sureda A, Andre M, Wahlin BE, Lugtenburg PJ, Jiang T, Karagoz K, Steele AJ, Abbas A, Wang L, Risum M, Cordoba R. Epcoritamab plus GemOx in transplant-ineligible relapsed/refractory DLBCL: results from the EPCORE NHL-2 trial. Blood. 2025 Apr 10;145(15):1621-1631. doi: 10.1182/blood.2024026830. PMID 39792928
- See also: Patient website: Recruiting clinical sites in Finland — https://fimea.fi/valvonta/kliiniset_laaketutkimukset/rekrytoivat-tutkimukset